CLINICAL TRIAL: NCT00589966
Title: Coping Skills Training Groups to Enhance Recovery From Prostate Cancer in African American Men
Brief Title: Coping in African American Prostate Cancer Survivors
Acronym: CAAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00000351; W81XWH-07-0091
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer treatment; treatment side-effects; early diagnosis; African American Men; coping skills training; quality of life; Prostate cancer treatment side-effects
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping Skills Training (Experimental)
  Interventions: Behavioral: Coping Skills Training
- Prostate Cancer Education (Active Comparator)
  Interventions: Behavioral: Prostate Cancer Education

INTERVENTIONS:
Behavioral: Coping Skills Training — Coping Skills Training teaches skills for managing physical, emotional, and social challenges of symptoms commonly experienced by men who have undergone treatment for early stage prostate cancer. Coping skills include activity pacing, managing negative mood, communication enhancement, and applied relaxation.
  Arms: Coping Skills Training
Behavioral: Prostate Cancer Education — Prostate Cancer Education provides information on the following topics: common treatment side-effects, medical options for symptom management, nutrition to support recovery, and guidelines for communicating with your healthcare team.
  Arms: Prostate Cancer Education

SUMMARY:
This study will test the effectiveness of an 8-week group intervention for African American men who have been treated for prostate cancer. The group intervention is based on 1) the cognitive-behavioral theoretical approach to improving adjustment to cancer and 2) masculinity theory as it relates to coping strengths and preferences in men. We will test the effectiveness of this coping skills intervention for improving survivors' quality of life in 4 areas: 1) distress related to sexual, urinary, and bowel symptoms; 2) self-confidence for managing symptoms; 3) overall emotional functioning; and 4) overall physical functioning. The effect of the coping skills group intervention in these 4 areas will be compared to a comparison intervention in which African American men will receive basic education about prostate cancer, but will not participate in coping skills training.

DETAILED DESCRIPTION:
African American men have higher diagnosis and death rates from prostate cancer than any other ethnic group. After treatment for prostate cancer, African American men also report slower recovery, including physical symptoms (e.g., sexual dysfunction, urinary incontinence) that can persist well beyond the immediate post-treatment period. Despite the evidence that African American men have poorer outcomes following prostate cancer treatment, very little is known about how to improve quality of life and enhance recovery in this group of survivors.

This study will test the effectiveness of an 8-week group intervention for African American men who have been treated for prostate cancer. The group intervention is based on 1) the cognitive-behavioral theoretical approach to improving adjustment to cancer and 2) masculinity theory as it relates to coping strengths and preferences in men. In this group intervention African American prostate cancer survivors will be taught a variety of coping skills for managing both the physical and emotional challenges of living with prostate cancer. The coping skills training groups will consist of 6-8 survivors and will be conducted in both medical center clinic settings and community settings (e.g., churches). Each group session will be co-led by an African American psychologist and an African American male lay person. We will test the effectiveness of this coping skills intervention for improving survivors' quality of life in 4 areas: 1) distress related to sexual, urinary, and bowel symptoms; 2) self-confidence for managing symptoms; 3) overall emotional functioning; and 4) overall physical functioning. The effect of the coping skills group intervention in these 4 areas will be compared to a comparison intervention in which African American men will receive basic education about prostate cancer, but will not participate in coping skills training. The recruitment goal for this project is 154 African American men treated for early stage prostate cancer.

Due to the comprehensive nature of the coping skills training intervention (i.e., a variety of coping skills targeting both physical and emotional challenges of prostate cancer), we expect coping skills training to be significantly more effective than cancer education. Ultimately, findings from this study could fill a significant gap that exists in the research literature regarding our understanding of how to help African American men achieve the fullest possible recovery following prostate cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early stage, localized prostate cancer (T1-T3)
* Must have received treatment within previous 2 years
* Capable of self-care per Karnofsky Performance Status score of 60+
* African American
* Must have physician who can confirm treatment history

Exclusion Criteria:

* Undergoing primary treatment 2 or more years ago
* Having regional or metastatic prostate cancer at time of screening

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Symptom distress | pretreatment, posttreatment, 3 mo followup

SECONDARY OUTCOMES:
Emotional functioning | pretreatment, posttreatment, 3 mo followup
Physical functioning | pretreatment, posttreatment, 3 mo followup
Self-efficacy for symptom management | pretreatment, posttreatment, 3 mo followup

CONTACTS AND LOCATIONS:
Overall Officials: Francis J Keefe, Ph.D., Principal Investigator — Duke University; Lisa C Campbell, Ph.D., Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States